CLINICAL TRIAL: NCT06546488
Title: Cognitive Assessment Tools for Individuals With Huntington's Disease.
Brief Title: Cognitive Assessment Tools for Huntington's Disease.
Acronym: CAT-HD
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Sandra Kostyk, Clinical Professor of Neurology, Ohio State University
Other Study IDs: 2024H0192
Record Dates: First submitted 2024-07-12; First posted 2024-08-09 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Huntington Disease
Keywords: Self-Administered Gerocognitive Examination (SAGE); Coding; Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject population: All subjects who meet the inclusion/exclusion criteria for the trial.
  Interventions: Behavioral: Assessments

INTERVENTIONS:
Behavioral: Assessments — A standardized assessment battery will be administered. It will consist of cognitive, functional and motor assessments.

SUMMARY:
The purpose of the current proposal is to expand understanding of two currently available cognitive tools that are not typically used in Huntington Disease (HD) clinical trials that might be useful both for initial screening and for clinical trial application. One is the Coding Test and the other is the Self-Administered Gerocognitive Examination (SAGE). Both the Coding Test and the SAGE have been used for assessments of individuals with other neurodegenerative diseases, including Alzheimer's Disease, Parkinson's Disease and Lewy Body Disease, but data is lacking on their use in individuals with HD.

DETAILED DESCRIPTION:
Subjects will be recruited from the OSU Wexner Medical Center Huntington Society of America Center of Excellence Clinic. Subjects will be scheduled for a one-time visit to complete the study. The entire visit will take approximately 1-1.5 hours. Vital signs (weight, blood pressure, temperature, respiratory rate and pulse) will be conducted. The subject's medical records will be reviewed to obtain their demographics, current medications, medical/surgical/ HD family history, and HD diagnosis details. If any adverse events occur during the research visit they will be documented. Participants will complete cognitive, functional and motor assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 30-65 (inclusive) at the time of signing the informed consent form.
2. Genetic diagnosis of HD as defined by a CAG repeat size ≥ 40.
3. A clinical diagnosis of HD as defined by a Diagnostic Confidence Level (DCL) of 4.
4. Vision and hearing sufficient for compliance with tests.
5. On a stable dose of medications for 30 days prior to the time of signing the informed consent form.

Exclusion Criteria:

1. Age of symptom onset less than 19 years old or greater than 60 years old.
2. Any serious neurological disorder aside from HD, including but not limited to Alzheimer's disease, Parkinson's disease, Frontotemporal dementia, Lewy body dementia, Amyotrophic Lateral Sclerosis, Traumatic Brain Injury… etc. that in the opinion of the investigator is clinically significant.
3. Any ongoing serious medical condition that in the opinion of the investigator is clinically significant. This includes autoimmune diseases, ongoing treatment for cancer, congestive heart failure, severe pulmonary disease, or any history of a seizure disorder (including the need to take anti-epileptics to prevent seizure).
4. Subjects who are pregnant or breast feeding
5. Subjects with a history of a learning disability.
6. Subjects who are unable to provide consent.

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Huntington disease patients with a clinical diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modality Test (SDMT) compared to the Coding Test | One day visit
  Comparison of scores on Symbol Digit Modality Test (SDMT) and Coding Test. Associations will be investigated using Spearman correlations.
Self-Administered Gerocognitive Examination (SAGE) score compared to the Symbol Digit Modality Test (SDMT) and the Stroop Word reading scores | One day visit
  Comparison of SAGE score with the SDMT and the Stroop Word reading scores. (The two neuropsychological scores used in the UHDRS that have shown the best correlation with HD disease onset and progression). Associations will be investigated using Spearman correlations.

SECONDARY OUTCOMES:
Comparison of Luria test scores and Symbol Digit Modality Test (SDMT) vs Coding scores. | One day visit
  Comparison of Luria test scores and SDMT vs coding scores. The Luria test is a sub-score of the Unified Huntington's Disease Rating Scale (UHDRS) motor exam and is considered marker of cognitive motor skill. Associations will be investigated using Spearman correlations.
Comparison of Total Motor Chorea sub-score, a part of the Unified Huntington's Disease Rating Scale (UHDRS) total score and scores on the Symbol Digit Modality Test (SDMT), Coding and Self-Administered Gerocognitive Examination (SAGE). | One day visit
  Comparison of Total Motor Chorea sub-score, a part of the UHDRS total score and scores on the SDMT, coding and SAGE.Severity of chorea involuntary movements that are common in HD might affect ability to complete either test as both the DSC and the SAGE require fine motor and drawing skills. Associations will be investigated using Spearman correlations.
Correlation of age of HD symptom onset and SAGE scores | One day visit
  Assess correlation of age of HD symptom onset and SAGE scores

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No